CLINICAL TRIAL: NCT07335406
Title: Registry for the Management of Helicobacter Pylori Infection in Shandong Province
Acronym: Hp-SHAREReg
Status: Not yet recruiting | Type: Observational
Sponsor: Yueyue Li (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Feicheng People's Hospital (Unknown); Binzhou Maternal and Child Health Hospital (Unknown); Jinxiang County People's Hospital (Unknown); The People's Hospital of Jimo (Unknown); Zibo Maternal and Child Health Hospital (Unknown); Yantai Penglai Traditional Chinese Medicine Hospital (Unknown); Zaozhuang Municipal Hospital (Other); Linyi Yizhou Hospital (Unknown); Taierzhuang District People's Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Yuncheng Traditional Chinese Medicine Hospital (Other); Caoxian County Hospital (Unknown); Qihe County People's Hospital (Unknown); University Town Hospital, Afiliated Hospital of Shandong University of Traditional Chinese Medicine (Unknown); Dezhou Hospital Qilu Hospital of Shandong University (Other); The 2nd People's Hospital of Dongying City (Unknown); Zhangdian District Hospital of Traditional Chinese Medicine (Unknown); Yantai Zhifu Hospital (Unknown); Inner Mongolia Autonomous Region International Mongolian Medicine Hospital (Unknown); Hohhot Second Hospital (Unknown); Guanxian People's Hospital (Unknown); Longkou People's Hospital (Unknown); Linshu County Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor-Investigator, Yueyue Li, Clinical Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: 202601
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Doctors prescribe Helicobacter pylori treatment regimens for patients based on current guidelines and consensus statements, tailored to individual circumstance, not involve any intervention procedure. — Doctors prescribe Helicobacter pylori treatment regimens for patients based on current guidelines and consensus statements, tailored to individual circumstance, not involve any intervention procedure.

SUMMARY:
Helicobacter pylori infection is a common global gastrointestinal infectious disease, affecting approximately 43.1% of the world's population. Eradicating H. pylori is crucial for reducing the risk of developing conditions such as gastritis, peptic ulcer disease, and gastric cancer. Currently, 14-day high-dose dual therapy containing amoxicillin and bismuth-containing quadruple therapy are the guideline-recommended first-line treatment regimens for H. pylori eradication. Treatment options for H. pylori vary considerably, with differing efficacy outcomes largely attributable to increasing bacterial antibiotic resistance. Furthermore, multiple factors influence the efficacy of H. pylori eradication, including smoking, body surface area, CYP2C19 gene polymorphisms, patient compliance, and regional variations.

Therefore, to systematically evaluate the efficacy and safety of different treatment regimens alongside the cost-effectiveness of various therapeutic strategies, and to conduct ongoing critical analysis of clinical practice, this study proposes a long-term investigation of real-world clinical practice through a non-interventional cohort study registry. This will assess the effectiveness, safety, and temporal trends of different H. pylori infection treatment regimens, providing real-time evidence to support clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-80 years, regardless of gender;
* willing to receive H. pylori eradication therapy;
* diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.

Exclusion Criteria:

* patients with incomplete medical records, including missing treatment details, absence of post-treatment follow-up test results, or failure to complete essential follow-up assessments;
* patients with severe underlying conditions such as hepatic insufficiency, renal insufficiency, or malignant tumours;
* pregnant or breastfeeding women;
* individuals who refuse to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) patients aged 18-80 years, regardless of gender; (2) willing to receive H. pylori eradication therapy; (3) diagnosed with H. pylori infection through at least one of the following methods: rapid urease test, ¹³C/¹⁴C-urea breath test, or histopathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2035-11-01 (Estimated); Study Completion 2035-11-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | at least 6 weeks after treatment completion

SECONDARY OUTCOMES:
Adverse events | lmmediately after treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China